CLINICAL TRIAL: NCT01261689
Title: The Randomised Epidural Analgesia in Term Delivering Women Trial
Brief Title: The Randomised Epidural Analgesia in Term Delivering Women Trial (TREAT)
Acronym: TREAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: TREAT01
Record Dates: First submitted 2010-11-10; First posted 2010-12-16 (Estimated); Last update posted 2013-11-27 (Estimated); Status verified 2013-11

CONDITIONS: Analgesia, Epidural; Instrumental Delivery; Maternal Outcome; Neonatal Outcome
Keywords: Epidural analgesia; Instrumental delivery; Maternal outcome; Neonatal outcome
MeSH Terms: conditions — Agnosia | interventions — Ropivacaine; Sufentanil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Epidural analgesia (Active Comparator): Women will be allocated to the EA group. In the EA group, women are given an EA as soon as they are in labour.
  Interventions: Drug: Ropivacaine/ Sufentanil according to local hospital protocol
- Care as-usual pain treatment (Other): Women will be allocated to the care-as-usual group. In this care-as-usual(restrictive) group, women receive pain relief only on their explicit request. If necessary epidural analgesia.
  Interventions: Other: Care-as usual pain treatment

INTERVENTIONS:
Drug: Ropivacaine/ Sufentanil according to local hospital protocol — according to local hospital protocol
  Other Names: ropivacaine/sufentanil
  Arms: Epidural analgesia
Other: Care-as usual pain treatment — Pain treatment only on request of the women in labour. Treatment is given according to local hospital protocol.
  Other Names: systemic opioids intramuscular and/or epidural analgesia
  Arms: Care as-usual pain treatment

SUMMARY:
* The objective of the study: to assess the impact of a proactive policy of offering EA at the start of labour as compared to a restrictive policy or care as usual.

* Study design: It concerns a multicentre randomised open label trial.

* Study population: Term nulliparous and multiparous women with a child in cephalic presentation, and without contraindications for vaginal labour or EA.

* Intervention: Women will be allocated to the EA group or the care-as-usual group. In the EA group, women are given an EA as soon as they are in labour. In the care-as-usual (restrictive) group, women receive pain relief only on their explicit request.

DETAILED DESCRIPTION:
Labour pain can be regarded as one of the most serious kinds of pain.In many countries labour pain is effectively treated on request of the labouring woman. In The Netherlands, labour pain has been traditionally approached conservatively. However, this policy is rapidly changing into effective treatments on request.Epidural analgesia (EA) has been proven to be one of the most effective methods of pain relief during labour.In addition, EA leads to increased patient satisfaction. Compared with other (or no) methods of pain relief, however, EA is associated with more use of oxytocin, a longer second stage of labour, and more instrumental vaginal deliveries. Other possible adverse effects in labouring women during EA are hypotension, motor block, urine retention, and fever. These complications and adverse effects are possible reasons, why EA is still not widely advised and accepted in The Netherlands.However, the question whether these adverse effects are caused by the EA, or that the observations are biased is still unanswered. The studies that have been performed to address these items are not applicable to the general population of women delivering a child, as they were all performed in women in strong need of pain relief.Generally, the need for pain relief is increased when progression of labour is difficult, for example in case of a relatively great child or ineffective contractions, especially in nulliparous women. It is well known that in this group of labouring women, also without EA, obstetrical problems are increased. On the other hand, a multivariable analysis of factors that are associated with an arrest of labour indicates, that women with EA have a decreased risk of arrest of labour. At present, randomized controlled trials that study the obstetrical consequences of EA in nulliparous women without strong need of pain relief are lacking. Besides that, only a few studies have extensively looked at the preference of women for EA. It seems that parity status, the fear of the side effects of EA, pain catastrophizing, the desire to have a pain-free childbirth, positive experiences with EA of family and friends influence the odds of choosing EA. So, based on the international literature, the ongoing increase in The Netherlands of EA's on maternal request during delivery may result in more obstetrical problems and increased health costs. Of course a change in pain treatment surrounding birth will have an impact for the women in labour, as well as for the society. On the one hand the costs of care are likely to increase due to EA, as EA is more expensive and might lead to an augmentation of medical complications, on the other hand in the EA-group women will have less pain while in labour as compared to the non-EA group. The question remains, whether this can be counteracted by a proactive policy of offering EA before explicit maternal request for pain relief in the absence of obstetrical problems. It is assumed, that a proactive policy might result in effective pain reduction and increased patient satisfaction without increased obstetrical problems and without increased health costs.

ELIGIBILITY:
Inclusion Criteria:

* be 18 years or older
* bear a singleton child in cephalic presentation
* be under supervision (second line) for their pregnancy in one of the participating centres.
* have no contraindications for vaginal labour
* have no contraindications for EA: Use of coumarines LMWH in therapeutic dose LMWH in prophylactic dose, less than 10 hours ago Thrombocytes < 80 x 109/ L Use of thrombocytes aggregation inhibitors or anamnestic increased bleeding tendency Blood clotting disorders Allergy for used anesthetics Spine disorders or back infection

Exclusion Criteria:

* be younger than 18 years
* bear twin pregnancy
* have contraindications for vaginal labour
* have contraindications for EA
* referral by midwife during labour (first line)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 488 (Actual)
Dates: Start 2008-09; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
instrumental delivery | at labour
  The primary outcome measure is the risk of an instrumental delivery (vaginal instrumental delivery and secondary cesarean sections)

SECONDARY OUTCOMES:
start labour | during labour
  start labour: spontaneous or induction
Oxytocin use | During labour
  Oxytocin use registration during labour.
Duration ruptured membranes | Labour
  Registration of duration of ruptured membranes
Internal digital vaginal examinations | Labour
  Counting of the total amount of vaginal examinations untill delivery
Maternal fever | During labour
  Defined as a temperature equal or above 38 degrees celsius.
Maternal antibiotic use | During labour
Duration of second stage of labour | labour
Obstetric complications | labour
  For example hemorrhagia postpartum defined as > 1000 ml or third/ fourt degree perinael rupture, shoulder dystocia.
Epidural related complications | labour and postpartum
  Epidural related complications, for example: bleeding, infection, postpunction headache.
Duration epidural | labour
  The duration in hours of the epidural untill the delivery.
Maternal hypotension | Labour
  Registration of the occurence of hypotension during labour.
Motor block | Labour
  Motor block defined by the brommage score (only patients with epidural)
Other use of anaesthetics | Labour
  Registration of the use of other used anaesthetics during labour.
Neonatal condition | Postpartum
  Apgar, umbilical blood gasses.
Neonatal antibiotic use | Postpartum
Neonatal admission | postpartum
Maternal pain catastrophizing | Antepartum
Beliefs about epidural | antepartum
  Inventarisation of the beliefs about epidural analgesia
Maternal childbirth experience | 6 weeks postpartum
  Inventarisation of the maternal childbirth experience
Quality of life | antepartum, 6 weeks postpartum
  Inventarisation of the quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Jan Nijhuis, Prof. MD, PhD, Study Chair — Maastricht University Medical Center; Martine Wassen, MD, Principal Investigator — Maastricht University Medical Center
Locations (2):
- Netherlands (2):
  - Atrium Medical Centre Parkstad, Heerlen, Limburg
  - Maastricht University Medical Centre, Maastricht, Limburg

REFERENCES:
- [Background] Wassen MM, Zuijlen J, Roumen FJ, Smits LJ, Marcus MA, Nijhuis JG. Early versus late epidural analgesia and risk of instrumental delivery in nulliparous women: a systematic review. BJOG. 2011 May;118(6):655-61. doi: 10.1111/j.1471-0528.2011.02906.x. Epub 2011 Mar 10. PMID 21392241